CLINICAL TRIAL: NCT02896946
Title: Use of Diffusion-weighted MRI for the Detection of Liver Metastases in Potentially Resectable Pancreatic Adenocarcinomas: a Prospective Multicenter Study
Brief Title: Diffusion MRI for Pancreatic Adenocarcinoma
Acronym: PANDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010.631
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2016-08

CONDITIONS: Pancreatic Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diffusion-weighted nuclear magnetic resonance imaging (Experimental): detection of liver metastasis on diffusion-weighted nuclear magnetic resonance imaging in patients with potentially resectable pancreatic adenocarcinoma
  Interventions: Radiation: Diffusion-weighted nuclear magnetic resonance imaging

INTERVENTIONS:
Radiation: Diffusion-weighted nuclear magnetic resonance imaging — All MRI examinations will be carried out using a Siemens Magnetom Avanto syngo MR B15 1.5 Tesla (Erlangen, Germany) or a Philips Intera 1.5 Tesla (Eindhoven, The Netherlands) and will include the following sequences: (i) T2 fat sat, with a FOV of 350 x 262, and a matrix of 384 x 207; slices, 30 per sequence, 6 mm thick; (ii) T1 in-phase and out-of-phase with a FOV of 380 x 262, and a matrix of 256 x 158; slices, 30 per sequence, 6 mm thick; (iii) T1 water excitation (= T1 ProSat), with a FOV of 300 x 300, and a matrix of 320 x 220; obtaining 20 slices of 4 mm; (iv) VIBE and THRIVE (dynamic T1 axial 3D EG after injection, during the arterial, portal venous, and late phases, in an axial plane, and optionally in a coronal plane during the portal venous phase), with a FOV of 400 x 312, a matrix of 384 x 192, and with fat suppression and breath-hold; slices 3 mm thick, with liver and pancreatic coverage. Contrast agent: gadobenate dimeglumine (MultiHance, Bracco Imaging, France).

SUMMARY:
The detection of small liver metastases represents a major challenge during the staging process of patients with pancreatic adenocarcinoma. Currently, thoraco-abdominopelvic CT represents the established imaging modality for selecting patients with pancreatic adenocarcinoma for curative surgery. However, despite its performance, 13% to 23% of patients undergoing a surgical procedure are finally found to have an unresectable disease because of arterial involvement, peritoneal carcinomatosis, or the existence liver metastasis that had not been detected by preoperative workup. Compared to CT, diffusion-weighted MRI provides a better contrast resolution for soft tissue and liver imaging, and thus leads to a better detection of focal liver lesions. Hence, it could be hypothesized that the use of DW-MRI in patients with potentially resectable PA may improve the selection process of candidates for curative pancreatic resection by increasing the detection of LM undiagnosed by traditional preoperative work-up

ELIGIBILITY:
Inclusion Criteria:

* age > 18 year old,
* no general contraindication for pancreatic surgery,
* pancreatic mass suspected or demonstrated to be a pancreatic adenocarcinoma,
* CAP CT of excellent technical quality showing a pancreatic tumor deemed resectable or border line (portal and/or superior mesenteric venous circumferential involvement < 180°
* Resectability confirmed by a medical/surgical multidisciplinary review,
* if neoadjuvant therapy was applied, patients were included in the study: only the second evaluation will be considered.
* informed consent prepared and signed.

Exclusion Criteria:

* locally advanced pancreatic adenocarcinoma (involvement > 180°in circumference of superior mesenteric venous (SMV) or portal vein, superficial vein thrombosis, superior mesenteric artery (SMA) involvement < 180°)
* unresectable tumour (circumferential involvement > 180 ° of the SMA, involvement of the celiac artery, thrombosis of the portal vein or vena cava, or complete VMS thrombosis
* metastasis of any organ visible on thoraco-abdominopelvic CT scan
* time lag exceeding 21 days between diffusion-weighted MRI and surgery
* contraindication for an MRI

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The rate of detection of liver metastasis on diffusion-weighted MRI in patients with potentially resectable pancreatic adenocarcinoma. | At the time of diagnosis of liver metastasis on histological study or based on follow-up (maximum time frame of 24 months after inclusion).
  The primary outcome will be measured at the time of diagnosis of liver metastasis, either based on histological study (within one month after surgery or biopsy) or based on follow-up (maximum time frame of 24 months after inclusion).

SECONDARY OUTCOMES:
Diagnostic performance of diffusion-weighted MRI for the preoperative diagnosis of liver metastasis in patients with potentially resectable adenocarcinoma | At the time of diagnosis of liver metastasis on histological study or based on follow-up (maximum time frame of 24 months after inclusion).
  Sensitivity, specificity, predictive positive value, negative predictive value and accuracy of diffusion-weighted MRI for the preoperative diagnosis of liver metastasis in patients with potentially resectable adenocarcinoma. The reference standard for the positive diagnosis of liver metastasis will be based on the pathological report of preoperative or intraoperative biopsies. In case of absence of tissue sample, the definitive diagnosis will be based on the 2-year follow-up.
Rate of patients for whom the therapeutic strategy is modified as a consequence of the diagnosis of liver metastasis on diffusion-weighted MRI | At the time of diagnosis of liver metastasis on histological study or based on follow-up (maximum time frame of 24 months after inclusion).
  Modification of therapeutic strategy is defined by abandonment of surgical exploration and/or of pancreatic excision after surgical exploration

REFERENCES:
- [Result] Marion-Audibert AM, Vullierme MP, Ronot M, Mabrut JY, Sauvanet A, Zins M, Cuilleron M, Sa-Cunha A, Levy P, Rode A. Routine MRI With DWI Sequences to Detect Liver Metastases in Patients With Potentially Resectable Pancreatic Ductal Carcinoma and Normal Liver CT: A Prospective Multicenter Study. AJR Am J Roentgenol. 2018 Nov;211(5):W217-W225. doi: 10.2214/AJR.18.19640. Epub 2018 Sep 21. PMID 30240298